CLINICAL TRIAL: NCT00001664
Title: Training Protocol for Various Sleep Disorders in Patients With Neurological Disorders
Brief Title: Sleep Disorders of Patients With Diseases of the Nervous System
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970070; 97-N-0070
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-07

CONDITIONS: Hypersomnia; Narcolepsy; Nervous System Disease; Sleep Disorder
Keywords: Narcolepsy; Polysomnography; Multiple Sleep Latency Test; Sleep Disorders; Hypersomnia; Periodic Leg Movements
MeSH Terms: conditions — Disorders of Excessive Somnolence; Narcolepsy; Nervous System Diseases; Sleep Wake Disorders

SUMMARY:
The purpose of this study is to assist training doctors about different diseases of the nervous system affecting sleep.

Patients selected to participate in this study will have any of a variety of sleep disorders. They will undergo several tests including an overnight recording of brain activity, eye movement, leg movement, breathing, heart rate, and other measures.

Results of these tests will be used to better understand diseases causing sleep disorders and may be used to develop better treatments for them.

DETAILED DESCRIPTION:
The objective of this protocol is to provide training in a broad range of neurological sleep disorders to clinical associates who are eligible for sitting in the Board examination of the Added Qualification of Clinical Neurophysiology administered by the American Board of Psychiatry and Neurology. This protocol is to supplement small accrual of research patients who are referred from within the NIH.

ELIGIBILITY:
* IINCLUSION CRITERIA:

Patients 5 years of age and older, with the following referring diagnoses:

Narcolepsy

Hypersomnia

REM behavior disorder

Frontal nocturnal dystonia

Restless legs syndrome

Insomnia

Parasomnia

Nocturnal epileptic seizure

Nocturnal movement disorder

Sleep-related diagnostic dilemma

Sleep apnea associated with neurological disorders

Patients who are ambulatory and who are able to comply with the study procedures.

Patients who are able to understand and sign the informed consent. (Parent or guardian for minors).

EXCLUSION CRITERIA:

Patients who have been diagnosed with acute and progressive neurological disorders.

Patients who are unable to comply with the study procedures and require other than standard care.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 1996-12-04; Study Completion 2011-09-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States